CLINICAL TRIAL: NCT00574275
Title: A Multinational, Randomized, Double-blind Study, Comparing the Efficacy of Aflibercept Once Every 2 Weeks Versus Placebo in Patients Treated With Gemcitabine for Metastatic Pancreatic Cancer
Brief Title: Aflibercept Compared to Placebo in Term of Efficacy in Patients Treated With Gemcitabine for Metastatic Pancreatic Cancer
Acronym: VANILLA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Data Monitoring Committee concluded after a planned interim analysis that aflibercept added to gemcitabine would be unable to demonstrate improved survival
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC10547; EudraCT 2007-003476-19
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Results first posted 2012-09-25 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-05

CONDITIONS: Pancreatic Neoplasm
Keywords: metastatic pancreatic cancer; angiogenesis inhibitor; gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — aflibercept; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo and Gemcitabine (Placebo Comparator): Participants with metastatic pancreatic cancer administered Placebo and 1000 mg/m^2 Gemcitabine.
  Interventions: Drug: Placebo; Drug: Gemcitabine
- Aflibercept and Gemcitabine (Experimental): Participants with metastatic pancreatic cancer administered 4 mg/kg Aflibercept and 1000 mg/m^2 Gemcitabine.
  Interventions: Drug: Aflibercept (ziv-aflibercept, AVE0005, VEGF trap, ZALTRAP®); Drug: Gemcitabine

INTERVENTIONS:
Drug: Aflibercept (ziv-aflibercept, AVE0005, VEGF trap, ZALTRAP®) — 4 mg/kg was administered intravenously (IV) over 1 hour once every 2 weeks, on Days 1 and 15 of each 28-day cycle.
  Arms: Aflibercept and Gemcitabine
Drug: Placebo — 4 mg/kg was administered intravenously (IV) over 1 hour once every 2 weeks, on Days 1 and 15 of each 28-day cycle
  Arms: Placebo and Gemcitabine
Drug: Gemcitabine — 1000 mg/m^2 administered IV over 30 minutes on Days 1, 8, 15, and 22 of Cycle 1 (28 days), and then Days 1, 8, and 15 of subsequent 28-day cycles.
  Other Names: Gemzar

SUMMARY:
The main objective of the study was to evaluate the effectiveness of aflibercept treatment by comparison to placebo in increasing the overall survival (OS) in participants with metastatic pancreatic cancer, treated with gemcitabine.

The secondary objectives were to evaluate progression free survival, clinical benefit, overall response, safety and immunogenicity of aflibercept, in the two treatment arms (Arm 1: Aflibercept and Gemcitabine; Arm 2: Placebo and Gemcitabine).

The study included an interim analysis of OS. In accordance with the study protocol, an interim analysis was performed for the purpose of futility and overwhelming efficacy. On the basis of the interim analysis, the Data Monitoring Committee (DMC) recommended that this study be terminated for futility based on predefined boundary rules.

DETAILED DESCRIPTION:
The study included:

* A screening visit of up to 21 days prior to randomization
* Randomization at baseline
* A Treatment period (initiated within 3 days of randomization), which included 28-day treatment cycles in both arms until predefined treatment discontinuation criteria were met
* A follow-up visit 30 days after discontinuation of treatment,
* A post study treatment follow-up period until death or the study cutoff date.

The criteria for treatment discontinuation were:

* Participant (or legal representative) chose to withdraw from treatment
* The investigator thought that continuation of the study would be detrimental to the participants well-being, such as:

  * Disease progression
  * Unacceptable AEs not manageable by symptomatic therapy, dose delay, or dose modification
  * Intercurrent illness that prevented further administration of study treatment
  * Noncompliance with the study protocol
* Participant was lost to follow-up
* Unblinding of the participant's investigational treatment

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically confirmed evidence of epithelial cancer (adenocarcinoma) of the exocrine pancreas
* Metastatic disease
* No prior chemotherapy for pancreatic disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Adequate renal, liver and bone marrow functions

Exclusion Criteria:

* Less than 42 days elapsed from prior major surgery (28 days from other prior surgery) to the time of randomization
* Prior treatment with anti-VEGF or VEGF-Receptor-inhibitors
* Uncontrolled hypertension
* Pregnancy or breastfeeding
* Participant with reproductive potential (M/F) without effective method of contraception

The above information is not intended to contain all considerations relevant to potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Actual)
Dates: Start 2007-12; Primary Completion 2009-10 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (24):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Sofia, Bulgaria
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Bogotá, Colombia
- Sanofi-Aventis Administrative Office, Nicosia, Cyprus
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Athens, Greece
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, San Juan, Puerto Rico
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Brastislava, Slovakia
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Geneva, Switzerland

REFERENCES:
- [Result] Rougier P, Riess H, Manges R, Karasek P, Humblet Y, Barone C, Santoro A, Assadourian S, Hatteville L, Philip PA. Randomised, placebo-controlled, double-blind, parallel-group phase III study evaluating aflibercept in patients receiving first-line treatment with gemcitabine for metastatic pancreatic cancer. Eur J Cancer. 2013 Aug;49(12):2633-42. doi: 10.1016/j.ejca.2013.04.002. Epub 2013 Apr 30. PMID 23642329

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between December 2007 and September 2009, a total of 546 participants were randomized in the study: 275 to the placebo group and 271 to the aflibercept group. On the basis of the interim analysis, the Data Monitoring Committee (DMC) recommended that this study be terminated for futility based on predefined boundary rules.
Groups:
- Placebo and Gemcitabine: * Placebo: 4 mg/kg was administered IV over 1 hour once every 2 weeks, on Days 1 and 15 of each 28-day cycle.
  * Gemcitabine: 1000 mg/m^2 administered IV over 30 minutes on Days 1, 8, 15, and 22 of Cycle 1 (28 days), and then Days 1, 8, and 15 of subsequent 28-day cycles.
- Aflibercept and Gemcitabine: * Aflibercept: 4 mg/kg was administered IV over 1 hour once every 2 weeks, on Days 1 and 15 of each 28-day cycle.
  * Gemcitabine: 1000 mg/m^2 administered IV over 30 minutes on Days 1, 8, 15, and 22 of Cycle 1 (28 days), and then Days 1, 8, and 15 of subsequent 28-day cycles.
Period: Overall Study
Arm/Group | Placebo and Gemcitabine | Aflibercept and Gemcitabine
Started | 275 | 271
TREATED | 273 | 268
SAFETY POPULATION | 271 (Excludes 2 participants who received 1 dose of Aflibercept) | 270 (Includes 2 participants from the Placebo and Gemcitabine arm who received 1 dose of Aflibercept)
Completed | 0 (All participants stopped when they met treatment discontinuation criteria or by DMC recommendation) | 0 (All participants stopped when they met treatment discontinuation criteria or by DMC recommendation)
Not Completed | 275 | 271
Not completed — Randomized but not treated | 2 | 3
Not completed — Adverse Event | 32 | 76
Not completed — Disease progression | 160 | 146
Not completed — Lost to Follow-up | 2 | 1
Not completed — Study stopped based on DMC decision | 62 | 23
Not completed — Withdrawal by Subject | 15 | 17
Not completed — Error calculating tumor measurement | 1 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Patient and Investigator decision | 0 | 1
Not completed — Insurance change | 0 | 1
Not completed — Operation for curative intent | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo/Gemcitabine: * Placebo: 4 mg/kg was administered IV over 1 hour once every 2 weeks, on Days 1 and 15 of each 28-day cycle.
  * Gemcitabine: 1000 mg/m^2 administered IV over 30 minutes on Days 1, 8, 15, and 22 of Cycle 1 (28 days), and then Days 1, 8, and 15 of subsequent 28-day cycles.
- Aflibercept/Gemcitabine: * Aflibercept: 4 mg/kg was administered IV over 1 hour once every 2 weeks, on Days 1 and 15 of each 28-day cycle.
  * Gemcitabine: 1000 mg/m^2 administered IV over 30 minutes on Days 1, 8, 15, and 22 of Cycle 1 (28 days), and then Days 1, 8, and 15 of subsequent 28-day cycles.
- Total: Total of all reporting groups
Arm/Group | Placebo/Gemcitabine | Aflibercept/Gemcitabine | Total
Number analyzed (Participants) | 275 | 271 | 546
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.4 (10.0) | 62.0 (9.4) | 61.2 (9.7)
Age, Customized [Number; unit: participants]
  <65 years | 179 | 161 | 340
  >=65 but <75 years | 77 | 90 | 167
  >=75 years | 19 | 20 | 39
Sex/Gender, Customized [Number; unit: participants]
  Male | 157 | 160 | 317
  Female | 118 | 111 | 229
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian/White | 267 | 256 | 523
  Black | 2 | 3 | 5
  Asian/Oriental | 3 | 7 | 10
  Other | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  ARGENTINA | 3 | 0 | 3
  AUSTRIA | 6 | 2 | 8
  BELGIUM | 18 | 16 | 34
  BULGARIA | 12 | 11 | 23
  CANADA | 15 | 16 | 31
  CHILE | 8 | 8 | 16
  CYPRUS | 3 | 3 | 6
  CZECH REPUBLIC | 10 | 14 | 24
  FRANCE | 11 | 13 | 24
  GERMANY | 15 | 10 | 25
  GREECE | 5 | 7 | 12
  HUNGARY | 7 | 10 | 17
  INDIA | 3 | 3 | 6
  ITALY | 17 | 24 | 41
  MEXICO | 1 | 2 | 3
  POLAND | 12 | 11 | 23
  PUERTO RICO | 1 | 0 | 1
  ROMANIA | 13 | 8 | 21
  RUSSIAN FEDERATION | 19 | 19 | 38
  SLOVAKIA | 5 | 3 | 8
  SPAIN | 13 | 14 | 27
  SWITZERLAND | 8 | 9 | 17
  UNITED STATES | 70 | 68 | 138
Eastern Cooperative Oncology Group (ECOG) Performance Status Score [Number; unit: participants] — The ECOG score assesses how the disease affects a participant's daily living abilities. It ranges from 0-5, with 0 being the best and 5 being the worst outcome. "0" reflects a fully active participant, able to carry on all pre-disease performance without restriction. "1" reflects a participant restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. "2" reflects an ambulatory participant, who is up and about more than 50% of waking hours, and capable of all self-care but unable to carry out any work activities.
  participants
    Participants with ECOG Score = 0 | 102 | 102 | 204
    Participants with ECOG Score = 1 | 154 | 152 | 306
    Participants with ECOG Score = 2 | 19 | 17 | 36
Primary tumor resection [Number; unit: participants] — Whether the participant had prior pancreatectomy.
  participants
    Yes | 40 | 39 | 79
    No | 235 | 232 | 467

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS is the time interval from the date of randomization to the date of death due to any cause. If death was not observed during the study, data on OS were censored at the earlier of the last date participant was known to be alive, or the study data cutoff date (11 September 2009).
  OS time was estimated from Kaplan-Meier Plots.
Time Frame: From the first randomization until the end of study data cutoff date (approximately 2 years)
Population: Intent-to-treat (ITT) population, which included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Units Other Than Participants: OS Event (Death)
Arm/Group | Placebo and Gemcitabine | Aflibercept and Gemcitabine
Number analyzed (Participants) | 275 | 271
Number analyzed (OS Event (Death)) | 142 | 142
months | 7.75 [6.768 to 8.575] | 6.54 [5.552 to 7.852]

2. Secondary Outcome: Progression Free Survival (PFS) Based on Response Evaluation Criteria in Solid Tumors [RECIST] Criteria
Description: PFS was the time interval from the date of registration to the date of progression, or death from any cause if it occurs before tumor progression is documented. Tumor progression was assessed using RECIST criteria, by which progression was a pre-defined increase in the size of existing tumors or appearance of one or more new tumors.
  If a participant did not progress or die, the progression was censored to the date of the last valid tumor assessment or data cut-off, whichever was earlier.
  Median PFS time was estimated from Kaplan-Meier Plots.
Time Frame: From the first randomization until the end of study data cutoff date (approximately 2 years)
Population: Intent-to-treat (ITT) population, which included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Units Other Than Participants: PFS Events
Arm/Group | Placebo and Gemcitabine | Aflibercept and Gemcitabine
Number analyzed (Participants) | 275 | 271
Number analyzed (PFS Events) | 189 | 182
months | 3.71 [3.515 to 4.567] | 3.71 [3.450 to 4.468]

3. Secondary Outcome: Objective Response Rate (ORR) Assessed by the Investigators According to RECIST Criteria
Description: Objective response (OR) included complete response [CR] and partial response [PR]. OR was to be assessed by the Investigators according to RECIST criteria, and confirmed by repeating tumor imaging at least 4 weeks after the first radiological documentation of response.
  CR would reflect the disappearance of all tumor lesions and PR would reflect a defined reduction of tumor burden.
  However, OR analysis was not performed, as the study was terminated due to futility.
Time Frame: From the first randomization until the end of the study data cutoff date (approximately 2 years)
Population: Since the study was terminated due to futility, this analysis was not performed.
Arm/Group | Placebo and Gemcitabine | Aflibercept and Gemcitabine
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Clinical Benefit
Description: Clinical benefit was to be assessed in all participants by time to symptom worsening (TTSW), evaluated from the time of randomization to symptom worsening, as well as by improvement in tumor related symptoms.
  However, this analysis was not performed, as the study was terminated due to futility.
Time Frame: From the first randomization until the end of the study data cutoff date (approximately 2 years)
Population: Since the study was terminated due to futility, analysis for this endpoint was not performed.
Arm/Group | Placebo and Gemcitabine | Aflibercept and Gemcitabine
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Safety-Number of Participants With Adverse Events (AE)
Description: All AEs regardless of seriousness or relationship to study treatment, spanning from the signature of informed consent until 30 days after the last administration of study treatment, were recorded. The number of participants with all treatment emergent adverse events (TEAE), serious adverse events (SAE), TEAE leading to death, and TEAE leading to permanent treatment discontinuation are reported.
Time Frame: up to 30 days after treatment discontinuation. SAEs and related AEs were followed till resolved or stabilized.
Population: The safety population included all randomized participants who were administered at least 1 dose of study medications (placebo, aflibercept, or gemcitabine). For safety analyses, participants were analyzed according to the treatment received.
Measure: Number; unit: participants
Arm/Group | Placebo and Gemcitabine | Aflibercept and Gemcitabine
Number analyzed (Participants) | 271 | 270
participants
  Treatment Emergent Adverse Event (TEAE) | 257 | 266
  Treatment Emergent Serious Adverse Event | 122 | 148
  TEAE leading to death | 43 | 55
  TEAE leading to permanent discontinuation | 32 | 76

6. Secondary Outcome: Number of Participants With Anti-drug Antibodies
Description: Anti-drug antibodies in the participants blood sample were detected using a validated immunoassay. The validated lower limit of detection (LLOD) for the assay was about 5.4 ng/mL in the absence of aflibercept and about 25.2 ng/mL in the presence of 20 μg/mL of aflibercept.
Time Frame: Up to 90 days post last dose of study drug
Population: Safety population with samples available for analysis
Measure: Number; unit: participants
Arm/Group | Placebo and Gemcitabine | Aflibercept and Gemcitabine
Number analyzed (Participants) | 202 | 201
participants | 5 | 5

ADVERSE EVENTS:
Time Frame: From treatment initiation up to November 26, 2010
Arm/Group | Placebo and Gemcitabine | Aflibercept and Gemcitabine
Serious Adverse Events (participants affected / at risk) | 122/271 | 148/270
Other Adverse Events (participants affected / at risk) | 239/271 | 249/270
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo and Gemcitabine (N=271) | Aflibercept and Gemcitabine (N=270)
Urinary tract infection (Infections and infestations) | 3 | 0
Pneumonia (Infections and infestations) | 3 | 2
Pharyngitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 2
Abdominal abscess (Infections and infestations) | 1 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Bacterascites (Infections and infestations) | 0 | 2
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 3 | 0
Biliary sepsis (Infections and infestations) | 2 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Peritoneal infection (Infections and infestations) | 0 | 1
Subdiaphragmatic abscess (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 2 | 0
Anal abscess (Infections and infestations) | 1 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0
Fungal oesophagitis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Splenic vein thrombosis (Blood and lymphatic system disorders) | 1 | 1
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 | 1
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 5 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Confusional state (Psychiatric disorders) | 0 | 2
Completed suicide (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 2 | 0
Syncope (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 2 | 1
Cerebellar syndrome (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Diabetic ketoacidotic hyperglycaemic coma (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 0
Monoplegia (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2
Cardiac failure (Cardiac disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Extrasystoles (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 4
Deep vein thrombosis (Vascular disorders) | 2 | 3
Thrombophlebitis superficial (Vascular disorders) | 1 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 2
Embolism arterial (Vascular disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 11 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 3
Vomiting (Gastrointestinal disorders) | 6 | 10
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 11 | 6
Stomatitis (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Ascites (Gastrointestinal disorders) | 2 | 4
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 4 | 4
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 4
Haematemesis (Gastrointestinal disorders) | 1 | 0
Duodenal obstruction (Gastrointestinal disorders) | 1 | 3
Duodenal stenosis (Gastrointestinal disorders) | 1 | 3
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 1
Melaena (Gastrointestinal disorders) | 0 | 2
Ileus (Gastrointestinal disorders) | 3 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Gastrointestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal oedema (Gastrointestinal disorders) | 1 | 0
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 2 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 3
Cholangitis (Hepatobiliary disorders) | 4 | 5
Bile duct obstruction (Hepatobiliary disorders) | 1 | 2
Bile duct stenosis (Hepatobiliary disorders) | 0 | 2
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 2
Cholangitis acute (Hepatobiliary disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 2 | 0
Hepatic failure (Hepatobiliary disorders) | 2 | 0
Portal hypertension (Hepatobiliary disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 2 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 2
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1
Epididymitis (Reproductive system and breast disorders) | 0 | 1
Fatigue (General disorders) | 5 | 1
Pyrexia (General disorders) | 5 | 3
Asthenia (General disorders) | 1 | 3
Disease progression (General disorders) | 25 | 38
Pain (General disorders) | 1 | 0
Device occlusion (General disorders) | 2 | 3
Performance status decreased (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Device dislocation (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Death (General disorders) | 4 | 0
Weight decreased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1
Blood glucose fluctuation (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo and Gemcitabine (N=271) | Aflibercept and Gemcitabine (N=270)
Urinary tract infection (Infections and infestations) | 17 | 16
Neutropenia (Blood and lymphatic system disorders) | 71 | 85
Thrombocytopenia (Blood and lymphatic system disorders) | 17 | 47
Decreased appetite (Metabolism and nutrition disorders) | 72 | 78
Insomnia (Psychiatric disorders) | 18 | 28
Depression (Psychiatric disorders) | 8 | 19
Anxiety (Psychiatric disorders) | 13 | 16
Headache (Nervous system disorders) | 19 | 51
Dysgeusia (Nervous system disorders) | 8 | 15
Hypertension (Vascular disorders) | 17 | 96
Deep vein thrombosis (Vascular disorders) | 16 | 9
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 | 40
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 37
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 14
Nausea (Gastrointestinal disorders) | 124 | 102
Vomiting (Gastrointestinal disorders) | 77 | 82
Diarrhoea (Gastrointestinal disorders) | 57 | 65
Constipation (Gastrointestinal disorders) | 73 | 64
Abdominal pain (Gastrointestinal disorders) | 61 | 54
Stomatitis (Gastrointestinal disorders) | 16 | 43
Abdominal pain upper (Gastrointestinal disorders) | 28 | 33
Rash (Skin and subcutaneous tissue disorders) | 19 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 23 | 27
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 14
Proteinuria (Renal and urinary disorders) | 6 | 30
Fatigue (General disorders) | 103 | 97
Pyrexia (General disorders) | 47 | 51
Asthenia (General disorders) | 42 | 51
Oedema peripheral (General disorders) | 43 | 33
Weight decreased (Investigations) | 43 | 81

LIMITATIONS AND CAVEATS:
As the study was terminated due to futility, some changes were made to the planned analyses, and the analyses for the following outcome measures were not performed:

* Objective Response Rate (ORR)
* Clinical Benefit

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to independently publish study results from his site after a multicenter publication, or 12 months after the completion of the study by all sites. He must provide the sponsor a copy of any such publication derived from the study for review and comment at least 45 days (20 days for abstracts) in advance of any submission, and delay publication till the approval of the publication is given in writing by the Sponsor (not to exceed ninety days).